CLINICAL TRIAL: NCT06096064
Title: Medication Use Evaluation (MUE) for Continuous Heparin Infusions in Hospitalized Patients
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 100.PHA.2022.R
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-09

CONDITIONS: Unfractionated Heparin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Unfractionated heparin (UFH) is an anticoagulant to prevent thrombus formation or worsening of an existing thrombus. It is indicated for patients with deep vein thrombosis/pulmonary embolism (DVT/PE) or acute coronary syndrome (ACS). Unfractionated heparin treatment consists of an initial bolus followed by a continuous infusion that is adjusted based on the patient's subsequent partial thromboplastin time (PTT) levels

DETAILED DESCRIPTION:
Unfractionated heparin is classified as a high-alert medication in the acute care setting.3 Therapeutic anticoagulation is a high priority for healthcare teams because the impacts of inadequate anticoagulation can lead to life threatening events such as a major bleed or thrombus formation and/or death.

ELIGIBILITY:
Inclusion Criteria:

* Patient's aged 18 years or older with a confirmed diagnosis of DVT/PE based on imaging or a confirmed diagnosis of ACS requiring heparin therapy

Exclusion Criteria:

* History of bleeding in the last 30 days
* History of HIT
* Use of systemic anticoagulants for another indication
* Presence of coagulation disorder prior to admission (i.e. hemophilia, sickle cell anemia, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: • Patient's aged 18 years or older with a confirmed diagnosis of DVT/PE based on imaging or a confirmed diagnosis of ACS requiring heparin therapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Incidents of deviations from protocol | 30 Days
  Appropriate anticoagulation management will be measured using Percent time in therapeutic range based on aPTT levels

CONTACTS AND LOCATIONS:
Locations (1):
- Methodist Richardson Medical Center, Dallas, Texas, United States